CLINICAL TRIAL: NCT02670629
Title: Management of Distal Radius Fractures in Children Younger Than 11 Years Old. Comparison Between Two Groups
Brief Title: Management of Distal Radius Fractures in Children Younger Than 11 Years Old.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carlos A Acosta-Olivo (Other)
Responsible Party: Sponsor-Investigator, Carlos A Acosta-Olivo, Professor - Orthopedics and Trauma Surgery, Universidad Autonoma de Nuevo Leon
Organization: Universidad Autonoma de Nuevo Leon (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OR14-011
Record Dates: First submitted 2016-01-22; First posted 2016-02-02 (Estimated); Results first posted 2019-11-14 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Bone Fractures; Radius Fractures; Closed Fractures
Keywords: Pediatric orthopedics
MeSH Terms: conditions — Fractures, Bone; Radius Fractures; Fractures, Closed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anatomic Closed Reduction + Short Cast (Active Comparator): Patients in this group were treated by performing a closed anatomic reduction under anesthesia by using sedatives and then placing the child in a short arm cast for 6 weeks. The follow up was done at week 1, 3, 6 and 10 with new X rays in each consult.
  The intervention in this control group was performing a closed anatomic reduction under anesthesia.
  Interventions: Procedure: Closed anatomic reduction
- Partial reduction overriding position (Experimental): Patients in this group were only given oral medications, the fracture was not reduced, instead it was left with a partial reduction with overriding position placed in a short arm cast for 6 weeks. The follow up was done at week 1, 3, 6 and 10 with new X rays in each consult.
  The intervention in this control group was not performing a closed anatomic reduction under anesthesia.
  Interventions: Procedure: Partial reduction with overriding position

INTERVENTIONS:
Procedure: Partial reduction with overriding position — The patient was subjected to an alignment instead of an anatomic reduction; this means that the fracture was left in an overriding position, after this, the patient was placed in a short arm cast for 6 weeks.
  Arms: Partial reduction overriding position
Procedure: Closed anatomic reduction — The patient was subjected to an anatomic reduction; this means that the fracture was completely reduced, after this, the patient was placed in a short arm cast for 6 weeks.
  Arms: Anatomic Closed Reduction + Short Cast

SUMMARY:
This fractures have been managed with anatomical reduction performed under anesthesia or using sedatives. In our institution this means prolonged hospital stay, involvement of an anesthesiologist and the use of an special room in the Emergency Department. This research protocol was born after reports were published regarding leaving the fractures in an overriding position and cast with good functional and acceptable radiographical results; said study was observational, providing valuable but limited information about this treatment option. On the other hand, our study is a randomized controlled trial between to groups of patients younger than 11 years old who presented to the Emergency Department with completely displaced distal radius fractures, they were randomly assigned to one of two groups, either a closed anatomic reduction and short cast or a closed overriding alignment and short cast.

DETAILED DESCRIPTION:
Distal radius fractures represent up to 40% of all fractures in pediatric patients, with the most common mechanism being simple falls with the hand and wrist in extension. The standard treatment for this kind of fractures is a closed anatomical reduction and placing a short arm cast for 6 week, with a weekly follow-up paying close attention to re-displacement and consolidation data. This fractures have acceptable deformity angles after the anatomical reduction of up to 15º in the coronal and sagittal plane; in order to perform this reduction, the patient is subject to a sedation under strict monitorization, either in the Emergency Department or in the Surgical Room. In most cases, the patient must stay in the hospital for at least 3 hours after the procedure was performed, in order to be discharged with analgesics and appropriate indications for caring a cast in home.

Distal radius fractures in pediatric patients have been managed with anatomical reduction performed under anesthesia or using sedatives. In our institution this means prolonged hospital stay, involvement of an anesthesiologist and the use of aa special room in the Emergency Department. This research protocol was born after reports were published regarding leaving the fractures in an overriding position and cast with good functional and acceptable radiographical results; said study was observational, providing valuable but limited information about this treatment option. On the other hand, our study is a randomized controlled trial between to groups of patients younger than 11 years old who presented to the Emergency Department with completely displaced distal radius fractures, they were randomly assigned to one of two groups, either a closed anatomic reduction and short cast or a closed overriding alignment and short cast.

Recent studies have suggested an alternative option for this patients, in which instead of performing a complete reduction, a gentle maneuver is done in order to get partial alignment or overriding fracture, with an strict follow-up and cooperative patients, this method has shown good results in terms of consolidation and deformity angles. The new procedure is performed without anesthesia, instead non-steroid antiinflammatory and analgesics are given to the patient, giving the possibility of an early discharge.

The possibility of leaving the patient with an overriding position and having good results is related to recent studies about bone in pediatric patients, especially in those younger than 14 years old. The published observations presume that fracture consolidation and remodeling potential is given by physis presence and the persistence throughout the years. Even more importantly, it is now known that the distal radius is predominantly formed by trabecular bone and a thicker periosteum, conditions that confer this bone a higher consolidation rate and rapid remodeling, leaving permanent deformities and reinterventions as rather rare situations. In terms of aesthetic deformities, 20º of radiological deformity in any plane is required to leave a clinically visible deformity, and even more so, 35º are needed to cause a functional impairment.

ELIGIBILITY:
Inclusion Criteria:

* Closed Completely displaced distal radius fractures with or without distal ulna fractures

Exclusion Criteria:

* Pathological Fractures
* Multiple Fractures
* Previous Fractures in either distal radius
* Metabolic Disease
* Open Fractures

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Fernando Mendoza Lemus, MD, PhD, Principal Investigator — Hospital Universitario José E Gonzalez

REFERENCES:
- [Background] Cannata G, De Maio F, Mancini F, Ippolito E. Physeal fractures of the distal radius and ulna: long-term prognosis. J Orthop Trauma. 2003 Mar;17(3):172-9; discussion 179-80. doi: 10.1097/00005131-200303000-00002. PMID 12621255
- [Result] Crawford SN, Lee LS, Izuka BH. Closed treatment of overriding distal radial fractures without reduction in children. J Bone Joint Surg Am. 2012 Feb 1;94(3):246-52. doi: 10.2106/JBJS.K.00163. PMID 22298057
- [Result] Friberg KS. Remodelling after distal forearm fractures in children. II. The final orientation of the distal and proximal epiphyseal plates of the radius. Acta Orthop Scand. 1979 Dec;50(6 Pt 2):731-9. doi: 10.3109/17453677908991303. PMID 532582
- [Result] Green JS, Williams SC, Finlay D, Harper WM. Distal forearm fractures in children:the role of radiographs during follow up. Injury. 1998 May;29(4):309-12. doi: 10.1016/s0020-1383(97)00208-8. PMID 9743754
- [Result] Hove LM, Brudvik C. Displaced paediatric fractures of the distal radius. Arch Orthop Trauma Surg. 2008 Jan;128(1):55-60. doi: 10.1007/s00402-007-0473-x. Epub 2007 Oct 17. PMID 17940779
- [Result] Pretell Mazzini J, Rodriguez Martin J. Paediatric forearm and distal radius fractures: risk factors and re-displacement--role of casting indices. Int Orthop. 2010 Mar;34(3):407-12. doi: 10.1007/s00264-009-0904-0. PMID 19916008
- [Result] Wilkins KE. Principles of fracture remodeling in children. Injury. 2005 Feb;36 Suppl 1:A3-11. doi: 10.1016/j.injury.2004.12.007. PMID 15652934
- Available data/document: Individual Participant Data Set: Fx radio distal — https://drive.google.com/open?id=0Bwd7ib0yn_zqMnBVZnY2NFFJTzA — Excel document with all the information regarding the patients included in this research protocol

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients in this research study were those admitted to the Emergency department of the Hospital Universitario "José Eleuterio González" between July 1, 2014 and December 1, 2015 with a diagnosis of a acute completely displaced distal radius fractures who matched our inclusion criteria.
Pre-assignment Details: Patients who had additional fractures or injuries, as well as those who sustained an open distal radius fractures were excluded from the trial before the assignment of groups. Other exclusion criteria included bone diseases, pathological fractures and chronic fractures.
Groups:
- Anatomic Closed Reduction + Short Cast: Patients in this group were treated by performing a closed anatomic reduction under anesthesia by using sedatives and then placing the child in a short arm cast for 6 weeks. The follow up was done at week 1, 3, 6 and 10 with new X rays in each consult.
  The intervention in this control group was performing a closed anatomic reduction under anesthesia.
  Closed anatomic reduction: The patient was subjected to an anatomic reduction; this means that the fracture was completely reduced, after this, the patient was placed in a short arm cast for 6 weeks.
- Partial Reduction Overriding Position: Patients in this group were only given oral medications, the fracture was not reduced, instead it was left with a partial reduction with overriding position placed in a short arm cast for 6 weeks. The follow up was done at week 1, 3, 6 and 10 with new X rays in each consult.
  The intervention in this control group was not performing a closed anatomic reduction under anesthesia.
  Partial reduction with overriding position: The patient was subjected to an alignment instead of an anatomic reduction; this means that the fracture was left in an overriding position, after this, the patient was placed in a short arm cast for 6 weeks.
Period: Overall Study
Arm/Group | Anatomic Closed Reduction + Short Cast | Partial Reduction Overriding Position
Started | 29 | 29
Completed | 29 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: We included 29 patients in both arms. All of the patients included in this trial completed the according follow-up.
Groups:
- Total: Total of all reporting groups
Arm/Group | Anatomic Closed Reduction + Short Cast | Partial Reduction Overriding Position | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.10 (2.05) | 8.59 (2.10) | 8.34 (2.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 11 | 15
  Male | 25 | 18 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 29 | 58
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Radial Shortening in Degrees - Residual Radiographic Deformities in Terms of the Radial Tilt, Radial Shortening and Radial Variation, Obtained in Both Groups.
Description: The cast was removed afer 6 weeks and rehabilitation in house was started as soon as the pain was over. The simple X rays were evaluated with the Montoya Classification, which stratifies the patients with regards of time until radiographic consolidation and bone remodeling. The radial tilt, radial shortening and radial variation was recorded and compared with the control group. This radiologic measures were reported in terms of degrees and millimeters were needed.
Time Frame: 10 weeks
Measure: Geometric Mean (Standard Deviation); unit: degrees
Arm/Group | Anatomic Closed Reduction + Short Cast | Partial Reduction Overriding Position
Number analyzed (Participants) | 29 | 29
degrees | 8.96 (1.2) | 8.998 (1.34)

2. Secondary Outcome: Pain Assessed by the Visual Analogue Scale (VAS) in Patients With Distal Radius Fractures Treated Without an Anatomical Reduction in Comparison to Those Treated With Anatomical Reduction.
Description: The Visual Analogue Scale (VAS) was used in order to assess the residual pain in the experimental group, this is, in patients with distal radius fractures treated without an anatomical reduction, this was later compared to the results obtained in the group in which a reduction was performed.
  Minimum value 0 maximum value 10. Higher score means a worse outcome.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anatomic Closed Reduction + Short Cast | Partial Reduction Overriding Position
Number analyzed (Participants) | 29 | 29
units on a scale | 3.4 (0.8) | 1.2 (0.7)

3. Secondary Outcome: Residual Functional Deficits Assessed by the UEFI (Upper Extremity Functional Index)in Patients With Distal Radius Fractures Treated Without an Anatomical Reduction.
Description: Patients were evaluated using a modified Upper Extremity Functional Index (UEFI) scale fot the appropriate age in order to assess functional deficits in the fractured limb in patients with distal radius fractures treated without an anatomical reduction.
  Evaluates the impairment the subject perceives they encounter when performing 20 types of activities of daily living. Each of the 20 actions in the UEFI is evaluated on a 5-point scale.
  Minimum Value 0 maximum value 4 per action, where 0 indicates most severe limitation and 80 suggests least limitation.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anatomic Closed Reduction + Short Cast | Partial Reduction Overriding Position
Number analyzed (Participants) | 29 | 29
units on a scale | 1.78 (0.062) | 0.755 (0.059)
Statistical Analysis 1: Comparison: Anatomic Closed Reduction + Short Cast vs Partial Reduction Overriding Position; Test type: Superiority or Other; p = 0.003, Chi-squared

4. Other Pre Specified Outcome: Aesthetic Results Measured by Clinical Radial Alignment in Degrees in Patients With Distal Radius Fractures Treated Without an Anatomical Reduction in Comparison to Those Treated With Anatomical Reduction in Both Groups.
Description: Patients were evaluated in comparison to the other extremity in terms of clinically evident deformity and appearance. Varus, Valgus, antecurvatum and recurvatum was measured and recorded appropriately. This was later compared to the data obtained in those patients who were treated with an anatomic reduction.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Anatomic Closed Reduction + Short Cast | Partial Reduction Overriding Position
Number analyzed (Participants) | 29 | 29
degrees
  Radius valgus | 2.5 (0.8) | 2.1 (0.7)
  Radius Varus | 2.1 (0.3) | 3.1 (0.5)
  Final Ulnar tilt | 1.2 (0.08) | 2.5 (1.2)

5. Primary Outcome: Patients With Residual Radiographic Deformities Obtained in Both Groups.
Description: as for outcome 1
Time Frame: 10 weeks
Measure: Number; unit: participants
Arm/Group | Anatomic Closed Reduction + Short Cast | Partial Reduction Overriding Position
Number analyzed (Participants) | 29 | 29
participants | 4 | 1

ADVERSE EVENTS:
Time Frame: The adverse event data was collected for 3 years.
Arm/Group | Anatomic Closed Reduction + Short Cast | Partial Reduction Overriding Position
Serious Adverse Events (participants affected / at risk) | 2/29 | 0/29
Other Adverse Events (participants affected / at risk) | 2/29 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anatomic Closed Reduction + Short Cast (N=29) | Partial Reduction Overriding Position (N=29)
Fracture redisplacement after reduction and cast (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — Two patients in our trial suffered a redisplacement after the fracture was reduced and placed in a cast. One o those patients needed a nail placed in the distal radius because of the fracture instability.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anatomic Closed Reduction + Short Cast (N=29) | Partial Reduction Overriding Position (N=29)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — One patient in our trial was left with residual pain and was managed with non steroid antiinflammatories.
Delayed Fracture Healing (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — One patient has a delayed fracture healing and was left in observation and protected with a sling for 6 weeks posterior to the cast.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No